CLINICAL TRIAL: NCT05195697
Title: ACUTE-Acute Surgical Care- Risk Factors and Outcomes for Patients in Need of Acute Surgical Care
Acronym: ACUTE
Status: Recruiting | Type: Observational
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-03583
Record Dates: First submitted 2022-01-04; First posted 2022-01-19 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Risk Factors; Complication of Surgical Procedure; Complication of Treatment; Complication of Anesthesia; Long Term Effects After Emergency Surgery; Long Term Effects After GI Bleeding
Keywords: Emergency surgery; Acute surgery; Complications; Risk factors; Frailty; Ageing
MeSH Terms: conditions — Frailty | interventions — Time-to-Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- Mild acute pancreatitis: Patients treated with mild acute pancreatitis during the study period
  Interventions: Other: Observational study of different treatments and time to treatment
- Moderate acute pancreatitis: Patients treated with moderate acute pancreatitis during the study period
  Interventions: Other: Observational study of different treatments and time to treatment
- Severe acute pancreatitis: Patients treated with severe acute pancreatitis during the study period
  Interventions: Other: Observational study of different treatments and time to treatment
- Acute gastrointestinal bleeding: Patients treated with acute gastrointestinal bleeding during the study period
  Interventions: Other: Observational study of different treatments and time to treatment
- Perforated ulcer: Patients treated with perforated ulcer during the study period
  Interventions: Other: Observational study of different treatments and time to treatment
- Older than 70 years: Patients older than 70 years
  Interventions: Other: Observational study of different treatments and time to treatment
- Less than 70 years: Patients younger than 70 years
  Interventions: Other: Observational study of different treatments and time to treatment
- Prothrombotic medications: Patients on prothrombotic medications
  Interventions: Other: Observational study of different treatments and time to treatment
- Frail patients: Patients with increased frailty score
  Interventions: Other: Observational study of different treatments and time to treatment
- Reintervention group: Patients in need of reintervention
  Interventions: Other: Observational study of different treatments and time to treatment

INTERVENTIONS:
Other: Observational study of different treatments and time to treatment — Different treatment based on the clinical decision

SUMMARY:
Observational retrospective study of patients in need of acute surgical care admitted to Skåne University Hospital between 2009 and 2019.

DETAILED DESCRIPTION:
At Skåne University Hospital approximately 6000 individuals are treated for acute abdominal diseases each year. Given the high number of patients, there is an urgent need to optimize acute surgical care. Lower complication rates would decrease hospital stay, health care costs as well as personal suffering.

Assessment instruments for risks and frailty are not validated for the acute setting and the investigators hypothesize there is room for improvement in prophylactic interventions and risk assessment. The investigators will study cohorts of patients with three different surgical diagnosis: acute pancreatitis, gastrointestinal bleeding and perforated ulcer aiming to identify risk factors for complications or death and to investigate assessment tools in this population. Using propensity score analysis, the investigators will try to identify treatment options associated with better outcome for subcohorts defined by frailty, comorbidity, age or gender. Specific factors of interest include: time to- and kind of treatment, handling of ongoing pharmacological therapy (anticoagulants, corticosteroids) and need for further treatments on a long time basis. The results from this project will be used in a future prospective study where prophylactic treatments and specific treatment options are studied.

ELIGIBILITY:
Inclusion Criteria: Patients admitted to Skåne University hospital in need of acute surgical care -

Exclusion Criteria: Below 18 years old

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients admitted to to Skåne University hospital in need of acute surgical care between 2009-2019
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | 5 years
  Defined by Swedish registers
Reintervention | 5 years
  Defined by medical records
Recurrent disease | 5 years
  Defined by medical records

SECONDARY OUTCOMES:
Lengths of hospital stay | 5 years
  defined by medical records
Number of interventions | 5 years
  defined by medical records
complications | 5 years
  defined by medical records and Swedish Registers

CONTACTS AND LOCATIONS:
Overall Officials: Sara Regnér, PhD, Principal Investigator — Region Skåne
Locations (1):
- Skåne University Hospital, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared after publication of studies from this trial upon request from publishers or other researchers. Only coded data will be shared and all sharing will be done according to the GDPR regulations.
Supporting Information: Study Protocol, SAP
Time Frame: Study protocol will be available during 2022. SAP will be available during 2023.
Access Criteria: After papers from this study have been published Upon request from publishers or researchers with a motivated scientific purpose or a motivated research question Only in accordance with GDPR regulations

REFERENCES:
- [Derived] Forsberg-Puckett A, Wurm Johansson G, Regner S. Presentation of gastrointestinal bleeding in patients with antithrombotic therapy, results from a consecutive retrospective cohort. Scand J Trauma Resusc Emerg Med. 2025 Sep 10;33(1):146. doi: 10.1186/s13049-025-01431-1. PMID 40931336